CLINICAL TRIAL: NCT04783168
Title: Ambulation to Improve Recovery With Wearable TECHnology (AIRTECH) Study
Brief Title: Walking After Surgery to Improve Recovery and Outcomes After Surgery, AIRTECH Study
Acronym: AIRTECH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-0453; NCI-2020-14126 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0453 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-02-03; First posted 2021-03-05 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Lung Carcinoma
Keywords: Wearable; device; fitness; tracker; Fitbit; ambulation; lung cancer; surgical; recovery
MeSH Terms: conditions — Lung Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Health Promotion; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm I (usual care) (Active Comparator): Patients receive usual care consisting of the clinician educating the patient on the importance of increasing exercise activity in the preoperative period and early ambulation in the postoperative setting.
  Interventions: Other: Best Practice; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (usual care, Fitbit) (Active Comparator): Patients receive usual care consisting of the clinician educating the patient on the importance of increasing exercise activity in the preoperative period and early ambulation in the postoperative setting. Patients also receive a Fitbit to monitor step count
  Interventions: Other: Best Practice; Other: Medical Device Usage and Evaluation; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm III (usual care, Fitbit, Fitbit app) (Experimental): Patients receive usual care consisting of the clinician educating the patient on the importance of increasing exercise activity in the preoperative period and walking in the postoperative setting. Patients also receive a Fitbit device, install and use the Fitbit app on a smartphone. Postoperative step goals are as follows: Postoperative day (POD) 1: 25% of baseline. Subsequent days will be increased by 10% until patient reaches baseline daily step number. Five automatic daily reminders (delivered by the Fitbit Inspire HR^TM device itself) to meet a minimum of 250 steps an hour. Postoperatively, patients will be invited to participate in a private group with a leaderboard that consists of step numbers of other participants in the study in an anonymous fashion.
  Interventions: Other: Best Practice; Other: Health Promotion and Education; Other: Medical Device Usage and Evaluation; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive usual care
  Other Names: standard of care; standard therapy
Other: Health Promotion and Education — Install and use Fitbit app
  Arms: Arm III (usual care, Fitbit, Fitbit app)
Other: Medical Device Usage and Evaluation — Use Fitbit to monitor step count
  Arms: Arm II (usual care, Fitbit); Arm III (usual care, Fitbit, Fitbit app)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial evaluates the relationship between walking and sleeping habits and surgical outcomes in patients with lung cancer. Early walking after surgery is associated with decreased or less severe complications. Learning about how much patients walk may be important in improving outcomes after surgery. Information gained from this trial may help researchers develop interventions to improve outcomes after surgery and improve overall quality of life after surgery in patients with lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Estimate the difference between each Fitbit arm and a control arm in Clavien-Dindo Combined Postoperative Morbidity (POM) Score in the 30-day postoperative period.

SECONDARY OBJECTIVES:

I. For patients in Fitbit only arm (F0) and Fitbit integration arm (FB), evaluate the differences in steps regained at each postoperative day.

II. Quality of life before and after surgery using MD Anderson Symptom Inventory - Lung Cancer (MDASI-LC).

III. Hospital length of stay. IV. Hospital readmission rate within 30 days for lung surgery related events. V. Return of bowel function. VI. Postoperative complications and step numbers. VII. Fitbit user experience in the FB arm.

EXPLORATORY OBJECTIVES:

I. Sleep disturbances. II. Cost analysis.

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM I: Patients receive usual care consisting of the clinician educating the patient on the importance of increasing exercise activity in the preoperative period and early ambulation in the postoperative setting.

ARM II: Patients receive usual care consisting of the clinician educating the patient on the importance of increasing exercise activity in the preoperative period and early ambulation in the postoperative setting. Patients also receive a Fitbit to monitor step count.

ARM III: Patients receive usual care consisting of the clinician educating the patient on the importance of increasing exercise activity in the preoperative period and walking in the postoperative setting. Patients also receive a Fitbit device install and use the Fitbit app on a smartphone. Postoperative step goals are as follows: Postoperative day (POD) 1: 25% of baseline. Subsequent days will be increased by 10% until patient reaches baseline daily step number. Five automatic daily reminders (delivered by the Fitbit Inspire HR^TM device itself) to meet a minimum of 250 steps an hour. Postoperatively, patients will be invited to participate in a private group with a leaderboard that consists of step numbers of other participants in the study in an anonymous fashion.

After completion of study intervention, patients are followed up at postoperative clinic and at 30 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* English speaking
* Ambulatory preoperatively
* Patients undergoing at least a lobectomy
* Must own a smart phone and be willing to install the Fitbit application (App)
* Adequate internet connection via wifi or wireless network connection with smartphone
* Patients who are not already using a wearable device to track daily steps

Exclusion Criteria:

* Medical, psychiatric, cognitive or other conditions that compromise the patient's ability to understand the patient information, to give informed consent, to comply with the study protocol or to complete the study.
* Cannot maintain activity monitor in place at the time of consent
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2020-11-30 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Clavien-Dindo postoperative morbidity (POM) score | Up to 30 days after surgery
  Two Bayesian probability and inferential models will be utilized:
  * Model 1: Inferential goals: Probability that POM score in the control arm is greater than F0 or FB arm: mean and 95% Credible Interval
  * Model 2: Baseline covariates adjusted analysis of model 1
    * Performance status
    * FEV1
    * Age
    * Open vs. Minimally invasive (0 is best, 5 is worst.) 0 - No postoperative complications 1. - Minor complication resolved without intervention 2. - complication requiring pharmaceutical intervention 3. - complication requiring surgical, endoscopic or radiological intervention, 4. - life-threatening complication requiring intensive care 5. - complication leading to the patient's death.

SECONDARY OUTCOMES:
Differences in steps regained at each postoperative day (Fitbit only arm [F0] and Fitbit integration arm [FB]) | Up to 30 days after surgery
  Number of steps regained starting from after surgery for each of the arms.
Change in quality of life | Baseline to 30 days after surgery
  Assessed using MD Anderson Symptom Inventory - Lung Cancer (MDASI-LC). (0 - 10 discrete numbers) 0 - Not present 10 - As bad as you can imagine.
Hospital length of stay | Up to 30 days after surgery
Hospital readmission rate for lung surgery related events | Up to 30 days after surgery
Return of bowel function | Up to 30 days after surgery
  Time to first bowel movement.
Postoperative complications and step numbers | Up to 30 days after surgery
  How would you rate daily step goals as being helpful in your postoperative recovery? From 0-5, 0 being not helpful at all and 5 being the most helpful.
Fitbit user experience (F0 and FB arm) | Up to 30 days after surgery
  Survey. How would you rate the use of Fitbit in your postoperative recovery From 0-5, 0 being not helpful at all and 5 being the most helpful How difficult was it to keep the device on your wrist From 0-5, 0 being extremely difficult, and 5 being extremely easy.

CONTACTS AND LOCATIONS:
Overall Officials: Garrett L Walsh, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org